CLINICAL TRIAL: NCT05495581
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ASP5354 in Participants With Renal Impairment Compared to Healthy Participants With Normal Renal Function
Brief Title: A Study About How ASP5354 Affects the Body in Healthy Adults and in Adults Whose Kidneys do Not Work Well
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5354-CL-0004
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers; Renal Impairment
Keywords: ASP5354; pudexacianinium chloride; Pharmacokinetics; Healthy Volunteers; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Mild renal impairment (Experimental): Participants will receive a single intravenous dose of ASP5354 under fasting conditions on Day 1.
  Interventions: Drug: pudexacianinium chloride
- Moderate renal impairment (Experimental): Participants will receive a single intravenous dose of ASP5354 under fasting conditions on Day 1.
  Interventions: Drug: pudexacianinium chloride
- Severe renal impairment (Experimental): Participants will receive a single intravenous dose of ASP5354 under fasting conditions on Day 1.
  Interventions: Drug: pudexacianinium chloride
- Normal renal function (Experimental): Participants will receive a single intravenous dose of ASP5354 under fasting conditions on Day 1.
  Interventions: Drug: pudexacianinium chloride

INTERVENTIONS:
Drug: pudexacianinium chloride — Intravenous
  Other Names: ASP5354

SUMMARY:
The ureter is the tube that carries urine from the kidneys to the bladder. It is difficult for surgeons to see the ureter during abdominal surgery. This could lead to injuring the ureter which, although rare, could be serious.

ASP5354 is a potential new medical dye to help surgeons clearly see the ureter during surgery. ASP5354 is injected into the body and is detected by a type of camera called near infrared fluoroscopy, or NIR-F for short. Together they show live images of the ureter during surgery.

Before ASP5354 is available as a medical dye, the researchers need to understand how it affects the body.

In this study, the researchers will check how ASP5354 affects the body in adults up to 75 years old. The main aim is to learn how ASP5354 is processed by the body in people whose kidneys do not work well compared to healthy people. There will be 4 groups of people with different levels of how well their kidneys work.

This study will include a 3-night stay in a clinical research unit. People will be admitted to the clinic the day before they receive the ASP5354 injection. The study doctor will take their medical history. People will have an ECG to measure their heart rhythm, a medical examination, and will have their vital signs checked (pulse rate, body temperature and blood pressure). They will also give blood and urine samples for laboratory tests. For some women, this will include a pregnancy test. People will need to fast for several hours before receiving the injection.

The next day, people will receive 1 injection of ASP5354. They will continue to fast for a few hours afterwards. They will have an ECG and will have their vital signs checked. They will also give blood and urine samples for laboratory tests and the study doctors will check for medical problems.

During the next 2 days, people will give more blood and urine samples and the study doctors will check for medical problems. On the last day, people will also have their vital signs checked. If there are no medical problems on the last day, people can return home.

People will return to the clinic about 1 week later for a final check-up. They will have an ECG, a medical examination and have their vital signs checked. They will give blood and urine samples for laboratory tests. For some women, this will include a pregnancy test. The study doctors will also check for medical problems.

ELIGIBILITY:
Inclusion Criteria:

For US study sites:

* Participant has a body mass index (BMI) range of 18.5 to 40.0 kg/m^2 inclusive and weighs at least 50 kg at screening.

For Japan study sites:

* Participant has a BMI range of 17.6 to 30.0 kg/m^2 inclusive and weighs at least 50 kg for male participants and 40 kg for female participants at screening.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of child bearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after study intervention administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 30 days after study intervention administration.
* Female participant must not donate ova starting at study intervention administration and throughout the study period and for 30 days after study intervention administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 30 days after study intervention administration.
* Male participant must not donate sperm during the treatment period and for 30 days after study intervention administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after study intervention administration.
* Participant agrees not to participate in another interventional study while participating in the present study.
* Participant has normal renal function or participant has varying degrees of chronic kidney disease (CKD) as defined by the National Kidney Foundation and calculated by individual estimated glomerular filtration rate (eGFR) using the modification of diet in renal disease (MDRD) formula and individual body surface area (BSA):

  * eGFR 60 to < 90 mL/min for participants with mild renal impairment
  * eGFR 30 to < 60 mL/min for participants with moderate renal impairment
  * eGFR < 30 mL/min without dialysis for participants with severe renal impairment, with approximately 50% of participants to have an eGFR of <= 20 mL/min
  * eGFR >= 90 mL/min for participants with normal renal function
* Participant has adequate venous access.

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half-lives whichever is longer, prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP5354, indocyanine green (ICG) or any components of the formulation used.
* Female participant who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Participant has had previous exposure with ASP5354.
* Participant has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST] and total bilirubin [TBL]) >= 1.5 x upper limit of normal [ULN] on day -1. In such a case, the assessment may be repeated once.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to study intervention administration.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Participant has a history of smoking > 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to day -1.
* For US study sites: Participant has a history of consuming > 14 units for male participants or 7 units for female participants of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1.
* For Japan study sties: Participant has a history of consuming > 16 units of alcohol per week within 3 months prior to day -1 (note: 1 unit = 10 grams pure alcohol, 250 ml of beer [5%], 35 milliliters [ml] of spirits [35%] or 100 ml of wine [12%]) or the participant tests positive for alcohol at screening or on day -1.
* For Japan study sites: Participant has body temperature < 35.0 degrees Celsius (C) or >= 37.5 degrees C on day -1.
* Participant has used any moderate or strong inducers of Cytochrome P450 family 3 subfamily A (CYP3A) in the 3 months prior to day -1.
* For US study sites: Participant has had significant blood loss, donated >= 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* For Japan study sites: Participant has had significant blood loss, donated >= 400 ml of whole blood within 90 days, >= 200 ml of whole blood within 30 days or donated blood components within 14 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* For US study sites: Participant has a positive serology test for hepatitis A Virus [HAV] antibodies (immunoglobulin M [IgM]), hepatitis B core [HBc] antibodies, hepatitis B surface antigen [HBsAg], hepatitis C virus [HCV] antibodies or antibodies to human immunodeficiency virus [HIV] type 1 and/or type 2 at screening.
* For Japan study sites: Participant has a positive serology test for HAV antibodies (IgM), HBc antibodies, HBsAg, HCV antibodies and/or antigen, antibodies to HIV type 1 and/or type 2 or syphilis at screening.
* Participant is an employee of Astellas, the study-related contract research organization (CRO) or the clinical unit.
* Participant has consumed grapefruit/Seville oranges or grapefruit/Seville orange-containing products within 72 hours prior to day -1.
* Participant has received a coronavirus disease 2019 (COVID-19) vaccine within the 2 weeks prior to study intervention administration or will have a COVID-19 vaccine dose before the end-of-study visit (ESV).
* Participant has a positive result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test at screening or on day -1.

Additional criteria for participants with renal impairment:

* Participant has a history of any clinically significant illness (other than renal disease and conditions related to the renal disease, such as stable diabetes and stable hypertension), medical condition or laboratory abnormality within 3 months prior to screening which preclude the participant from study participation.
* For US study sites: Participant has a mean pulse < 40 or > 90 beats per minute (bpm); mean systolic blood pressure (SBP) < 90 or > 160 mmHg; mean diastolic blood pressure (DBP) < 50 or > 100 millimeters mercury [mmHg] (measurements taken in triplicate after the participant has been resting in a supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* For Japan study sites: Participant has a mean pulse < 40 or > 90 bpm; mean SBP < 90 or > 160 mmHg; mean DBP < 40 or > 90 mmHg (measurements taken in triplicate after the participant has been resting in a supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* For US study sites: Participant has a mean corrected QT interval by Fridericia (QTcF) of > 450 msec for male participants and > 480 msec for female participants on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate electrocardiogram (ECG) may be taken.
* For Japan study sites: Participant has a mean QTcF of > 450 msec for male participants and > 470 msec for female participants on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant who has had a change in dose regimen of medically required medication(s) in the 2 weeks prior to study intervention administration (permitted concomitant medications) and/or participant for whom dose changes are likely to occur during the study (minor dose changes are allowed in agreement with the sponsor) and/or participant has used nonpermitted concomitant medication(s) in the 3 weeks prior to admission to the clinical unit.
* Participant who requires or is likely to require any new concomitant medications during the course of the study.
* Participant who has a renal disease secondary to malignancy.
* Participant who has a fluctuating or rapidly deteriorating renal function within 4 weeks prior to study intervention administration, as indicated by strongly varying or worsening of clinical and/or laboratory signs of renal impairment within the screening period.
* Participant has a hemoglobin result of < 9 grams/deciliter (g/dL).
* Participant has a functioning kidney transplant.
* For US study sites: Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on day -1, unless the positive result is due to an approved prescription medication.
* For Japan study sites: Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or morphine, phencyclidines and tricyclic antidepressants) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or morphine, phencyclidines and tricyclic antidepressants) at screening or on day -1, unless the positive result is due to an approved prescription medication.

Additional criteria for healthy participants with normal renal function:

* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has any clinically significant abnormality following the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1.
* For US study sites: Participant has a mean pulse < 45 or > 90 bpm; mean SBP > 140 mmHg; mean DBP > 90 mmHg (measurements taken in triplicate after the participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* For Japan study sites: Participant has a mean pulse < 40 or > 100 bpm; mean SBP < 90 or > 140 mmHg; mean DBP < 40 or > 90 mmHg (measurements taken in triplicate after the participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean QTcF of > 450 msec for both male and female participants on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study intervention administration, except for occasional use of acetaminophen (up to 2 grams/day), topical dermatological products (including corticosteroid products), hormonal contraceptives and hormone replacement therapy (HRT).
* Participant has creatinine level outside normal limits on day -1. In such a case, the assessment may be repeated once.
* For US study sites: Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on day -1.
* For Japan study sites: Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or morphine, phencyclidines and tricyclic antidepressants) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or morphine, phencyclidines and tricyclic antidepressants) at screening or on day -1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of ASP5354 in plasma: area under the concentration-time curve from time of dosing extrapolated to time infinity (AUCinf) | Up to 3 days
  AUCinf will be recorded from the pharmacokinetic (PK) plasma samples collected.
PK of ASP5354 in plasma: area under concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Up to 3 days
  AUClast will be recorded from the pharmacokinetic (PK) plasma samples collected.
PK of ASP5354 in plasma: maximum concentration (Cmax) | Up to 3 days
  Cmax will be recorded from the pharmacokinetic (PK) plasma samples collected.
PK of ASP5354 in plasma: apparent clearance (CL) | Up to 3 days
  CL will be recorded from the pharmacokinetic (PK) plasma samples collected.
PK of ASP5354 in urine: cumulative amount of unchanged drug excreted in urine from time of dosing to time infinity after single dose (Aeinf) | Up to 3 days
  Aeinf will be recorded from the pharmacokinetic (PK) urine samples collected.
PK of ASP5354 in urine: cumulative amount of unchanged drug excreted in urine from time of dosing to the last measurable amount (Aelast) | Up to 3 days
  Aelast will be recorded from the pharmacokinetic (PK) urine samples collected.
PK of ASP5354 in urine: cumulative amount of unchanged drug excreted in urine from time of dosing to time infinity after single dose as a percentage of total cumulative amount of unchanged drug excreted in urine (Aeinf%) | Up to 3 days
  Aeinf% will be recorded from the pharmacokinetic (PK) urine samples collected.
PK of ASP5354 in urine: cumulative amount of unchanged drug excreted in urine from time of dosing to the last measurable amount as a percentage of total cumulative amount of unchanged drug excreted in urine (Aelast%) | Up to 3 days
  Aelast% will be recorded from the pharmacokinetic (PK) urine samples collected.
PK of ASP5354 in urine: renal clearance (CLr) | Up to 3 days
  CLr will be recorded from the pharmacokinetic (PK) urine samples collected.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 12 days
  AEs will be coded by Medical Dictionary for Regulatory Activities (MedDRA). An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  Note: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator and events related to the (study) procedures.
Number of participants with laboratory value abnomalities and/or AEs | Up to 12 days
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital signs abnormalities and/or AEs | Up to 12 days
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 12 days
  Number of participants with potentially clinically significant ECG values.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- United States (3):
  - Pinnacle Research Group, Anniston, Alabama
  - Orange County Research Center, Tustin, California
  - Advanced Pharma CR, LLC, Miami, Florida
- Sekino Clinical Pharmacology Clinic, Toshima-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.